CLINICAL TRIAL: NCT06582355
Title: MOTOR-NF - a Randomized Controlled Trial of FMRI-based Neurofeedback for Motor Symptoms of Parkinson's Disease
Brief Title: FMRI-neurofeedback in Parkinson's Disease
Acronym: MOTOR-NF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL86308.068.24
Record Dates: First submitted 2024-05-06; First posted 2024-09-03 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Neurofeedback; fMRI
MeSH Terms: conditions — Parkinson Disease | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware of which condition the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurofeedback (Experimental): Four weekly MRI sessions where they will learn to upregulate the activity of the putamen during motor imagery via fMRI neurofeedback.
  Interventions: Other: Neurofeedback
- Kinesthetic imagery (Active Comparator): Four weekly MRI sessions with motor imagery without fMRI neurofeedback.
  Interventions: Other: Kinesthetic imagery

INTERVENTIONS:
Other: Neurofeedback — The participants will be instructed to use cognitive strategies to upregulate (increase) their brain activity in the selected brain region, with the suggestion that motor imagery may be particularly effective, for example, mental imagery of swimming or playing a musical instrument. During the rest blocks, the participants will be instructed to relax. The instructions to start and stop the regulation and rest blocks are visualized on a screen in the scanner, and the brain activity of the putamen will be displayed in real-time using a thermometer bar for visualization.
  Arms: Neurofeedback
Other: Kinesthetic imagery — The participants will be instructed to imagine movements during the active blocks. During the rest blocks, the participants will be instructed to relax. The instructions to start and stop the regulation and rest blocks are visualized on a screen in the scanner. No feedback is provided regarding brain activity.
  Arms: Kinesthetic imagery

SUMMARY:
Rationale: Current treatment of patients with Parkinson's disease (PD) is mainly based on the modulation of neural activity in the motor circuits of the basal ganglia and cerebral cortex by either drug intervention (dopamine replacement therapy or dopaminergic medication) or deep brain stimulation (DBS). However, many Parkinson patients have an insufficient (long-term) response to medical treatments, and DBS is an invasive procedure with resource implications and potential side effects. Moreover, not all patients are eligible for DBS. Therefore, new ways of administering neuromodulation are needed. A potential avenue may be self-regulation of brain circuits through neurofeedback. Self-regulation of motor circuits through mental imagery and neurofeedback using real-time functional MRI (fMRI) signals has already been shown to be feasible, and there are also preliminary data on clinical benefits of such self-regulation training. We here aim to use the non-invasive fMRI-neurofeedback method to train patients in the regulation of brain circuits that are implicated in successful drug treatment and/or DBS.

Objective: To investigate brain mechanisms and efficacy of an fMRI-neurofeedback protocol that targets the brain's motor circuits through the basal ganglia.

Study design: Randomised controlled trial Study population: Patients with Parkinson's disease Investigation: In the experimental group, fMRI-neurofeedback will be administered in 4 separate sessions of about 2 hours each over approximately one month. The MRI measurement in each session will be approximately 60 minutes long and include upregulation training of brain activity in specific target areas by mental imagery. The fMRI signals are processed such that the patients get visual feedback about the success of the upregulation. In addition, patients are asked to practice the self-regulation strategies on a daily basis at home between the neurofeedback sessions. The control intervention will consist of mental imagery without neurofeedback.

Main study parameters/endpoints: Post-interventional improvement of motor symptoms of PD as assessed by the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) motor scale in the on-medication state.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This is a low-risk study where the main burden is participation time and MRI scans.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is associated with progressive neurodegeneration of dopaminergic neurons of the substantia nigra. It is characterized by both motor and non-motor system manifestations. Dopamine replacement therapy or dopaminergic medication are the key therapeutic strategies, but deep brain stimulation (DBS) is increasingly being used in cases where drug response is/ has become insufficient or hampered by unacceptable side effects.

Neurofeedback (NF) entails training of self-regulation of brain regions or networks via mental imagery and real-time feedback of neural signals, for example obtained by functional MRI (fMRI). NF enables patients to develop personal strategies that are most effective in self-regulating brain areas and networks. Thereby, it can provide an individually tailored intervention. NF is a highly sustainable form of non-invasive neuromodulation because, once learnt, the self-regulation strategies can in principle be applied by patients whenever needed to overcome disease symptomology.

NF can be used to train patients to change their brain activity in different directions, or to modulate patterns of co-activation between regions. Mental imagery of moving one's own body (also called kinaesthetic imagery) can potentially be used to improve motor functions and neuroplasticity in PD. Kinaesthetic imagery is also a suitable strategy for increasing activation in the brain's motor network, and motor imagery training can be reinforced through combination with NF. A NF paradigm involving upregulation training of motor areas through kinaesthetic imagery thus has good plausibility for PD. The PI's group has shown proof-of-concept of such an fMRI-NF training (targeting the supplementary motor area, SMA) in PD and has recently completed a feasibility study of fMRI-NF targeting the putamen in 12 PD patients (NCT05627895). The aim of the current investigator-initiated study is to investigate the effects of putamen upregulation training on motor function and other outcome parameters in PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease.
* Disease stage 1-3 according to the Hoehn and Yahr Scale
* Age: 18 years or more

Exclusion Criteria:

* Exclusion criteria for MRI (e.g., cardiac pacemaker, certain metallic implants)
* History of psychotic disorder, bipolar disorder, or psychotic depression
* Current use of illegal drugs (any in the last four weeks)
* Current excessive alcohol consumption that interferes with daily functioning
* A score on the Montreal Cognitive Assessment (MoCA) below 24/30.
* Any disorder that would interfere with accurate and usable data acquisition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS (Unified Parkinson's Disease Rating Scale) | After screening, after the last MRI session (approx. 5 weeks after screening) and at follow up session (approx. 4 weeks after final MRI session)
  Pre versus Post-interventional change in the MDS-UPDRS (Unified Parkinson's Disease Rating Scale) motor scale will be compared using t statistics.
  The MDS-UPDRS contains 65 scores, each with a range from 0 (no impairment) to 4 (severe impairment).
  The total scale ranges between 0 - 260, with 0 indicating no impairment and 260 indicating the highest level of impairment.
  As primary outcome measure we will use Part III: Motor Examination, which has 33 scores. The measurement at the last MRI session will be the primary endpoint.

SECONDARY OUTCOMES:
Performance of Putamen neurofeedback training (fMRI analysis) | Measurements will be recorded at each MRI session (approx. 1 week intervals after screening and inclusion)
  To determine the performance of Putamen self-regulation, we will employ an region of interest (ROI) general linear model analysis, using a T-contrast of all blocks with the Putamen as the target region versus all the baseline blocks. This will allow us to assess recruitment of the Putamen during the training as well as regulation success.
  Furthermore we will use an ANOVA F-contrast to check for any interactions of the neurofeedback training with sessions (eg., if Session 4 shows improved neurofeedback success as compared to Session 1).
Whole brain activation pattern changes (fMRI analysis) | Measurements will be recorded at each MRI session (approx. 1 week intervals after screening and inclusion)
  We will investigate the whole brain level activation pattern changes due to neurofeedback training using self-regulation in PD patients. To determine these changes, we will look at the T-contrast of all regulation blocks vs all baseline blocks in all the fMRI runs with neurofeedback. This can give us insight into which brain networks contribute mechanistically to the training and if any of the training performance can be attributed to other factors, such as physiological measures, as compared to neurofeedback self-regulation.
Neurofeedback training effects on non-motor symptoms | After screening, after the last MRI session (approx. 5 weeks after screening) and at follow up session (approx. 4 weeks after final MRI session)
  Effect of neurofeedback training on non-motor symptoms will be assessed using the MDS-UPDRS part I, II, IV and the Hospital Anxiety and Depression Scale (HADS).
  The MDS-UPDRS contains 65 scores, each with a range from 0 (no impairment) to 4 (severe impairment).
  The Part I subscore, indicating nonmotor experiences of daily living has a total of 13 items with scores ranging between 0-52.
  The HADS is a widely used questionnaire designed to assess levels of anxiety and depression in patients. It consists of 14 items, with seven questions related to anxiety (HADS-A) and seven related to depression (HADS-D). Each item is scored on a scale from 0 to 3, with total scores ranging from 0 to 21 for each subscale. The HADS is commonly used in clinical settings to identify and measure the severity of anxiety and depression in patients, particularly in hospital environments.
Correlation between NF success and distal finger tapping test (behavioral measure) | After screening, after the last MRI session (approx. 5 weeks after screening) and at follow up session (approx. 4 weeks after final MRI session)
  We will correlate neurofeedback success with the distal finger tapping (DFT) test scores to determine if NF success can lead to improvements in behavioral measures.
  Three kinetic parameters are generated by the DFT test: kinesia score (KS20), the number of keystrokes in a 20 second time period, reflecting speed; akinesia time (AT20), average dwell time that keys are depressed, reflecting akinesia; and incoordination score (IS20), the variance of travelling time between keystrokes, reflecting rhythm. A higher KS20 score represents improvement, a lower AT20 score represents improvement and a smaller variance in the IS20 score represents improvement.

OTHER OUTCOMES:
Neurofeedback training effects on motor symptoms and experiences | After screening, after the last MRI session (approx. 5 weeks after screening) and at follow up session (approx. 4 weeks after final MRI session)
  Effect of neurofeedback training on motor symptoms and experiences will be assessed using the MDS-UPDRS part II and IV.
  The MDS-UPDRS contains 65 scores, each with a range from 0 (no impairment) to 4 (severe impairment).
  The Part II subscore, indicating nonmotor experiences of daily living has a total of 13 items with scores ranging between 0-52.
  The Part IV subscore, indicating nonmotor experiences of daily living has a total of 6 items with scores ranging between 0-24.

CONTACTS AND LOCATIONS:
Overall Officials: David EJ Linden, Prof., Principal Investigator — Maastricht University
Locations (2):
- Uniklinik Köln, Cologne, Germany
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akram N, Li H, Ben-Joseph A, Budu C, Gallagher DA, Bestwick JP, Schrag A, Noyce AJ, Simonet C. Developing and assessing a new web-based tapping test for measuring distal movement in Parkinson's disease: a Distal Finger Tapping test. Sci Rep. 2022 Jan 10;12(1):386. doi: 10.1038/s41598-021-03563-7. PMID 35013372
- [Background] Emmert K, Kopel R, Sulzer J, Bruhl AB, Berman BD, Linden DEJ, Horovitz SG, Breimhorst M, Caria A, Frank S, Johnston S, Long Z, Paret C, Robineau F, Veit R, Bartsch A, Beckmann CF, Van De Ville D, Haller S. Meta-analysis of real-time fMRI neurofeedback studies using individual participant data: How is brain regulation mediated? Neuroimage. 2016 Jan 1;124(Pt A):806-812. doi: 10.1016/j.neuroimage.2015.09.042. Epub 2015 Sep 28. PMID 26419389
- [Background] Esmail, S., & Linden, D. E. J. (2014). Neural Networks and Neurofeedback in Parkinson's Disease. NeuroRegulation, 1(3-4), 240-240. https://doi.org/10.15540/nr.1.3-4.240
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Hamilton JP, Glover GH, Bagarinao E, Chang C, Mackey S, Sacchet MD, Gotlib IH. Effects of salience-network-node neurofeedback training on affective biases in major depressive disorder. Psychiatry Res Neuroimaging. 2016 Mar 30;249:91-6. doi: 10.1016/j.pscychresns.2016.01.016. Epub 2016 Jan 19. PMID 26862057
- [Background] Jaeckle T, Williams SCR, Barker GJ, Basilio R, Carr E, Goldsmith K, Colasanti A, Giampietro V, Cleare A, Young AH, Moll J, Zahn R. Self-blame in major depression: a randomised pilot trial comparing fMRI neurofeedback with self-guided psychological strategies. Psychol Med. 2023 May;53(7):2831-2841. doi: 10.1017/S0033291721004797. Epub 2021 Dec 2. PMID 34852855
- [Background] Johnston SJ, Boehm SG, Healy D, Goebel R, Linden DE. Neurofeedback: A promising tool for the self-regulation of emotion networks. Neuroimage. 2010 Jan 1;49(1):1066-72. doi: 10.1016/j.neuroimage.2009.07.056. Epub 2009 Jul 29. PMID 19646532
- [Background] Karch, S., Keeser, D., Paolini, M., Hümmer, S., Konrad, J., Haller, D., Kirsch, V., Koller, G., Kupka, M., Blautzik, J., & Pogarell, O. (2015). Real-time fMRI neurofeedback: Applica-tion in patients with substance use disorder. Pharmacopsychiatry, 25(6), A77. https://doi.org/10.1055/s-0035-1558015
- [Background] Linden DE. Neurofeedback and networks of depression. Dialogues Clin Neurosci. 2014 Mar;16(1):103-12. doi: 10.31887/DCNS.2014.16.1/dlinden. PMID 24733975
- [Background] Linden DE, Habes I, Johnston SJ, Linden S, Tatineni R, Subramanian L, Sorger B, Healy D, Goebel R. Real-time self-regulation of emotion networks in patients with depression. PLoS One. 2012;7(6):e38115. doi: 10.1371/journal.pone.0038115. Epub 2012 Jun 4. PMID 22675513
- [Background] MacDuffie KE, MacInnes J, Dickerson KC, Eddington KM, Strauman TJ, Adcock RA. Single session real-time fMRI neurofeedback has a lasting impact on cognitive behavioral therapy strategies. Neuroimage Clin. 2018 Jun 9;19:868-875. doi: 10.1016/j.nicl.2018.06.009. eCollection 2018. PMID 29922575
- [Background] Mehler DMA, Sokunbi MO, Habes I, Barawi K, Subramanian L, Range M, Evans J, Hood K, Luhrs M, Keedwell P, Goebel R, Linden DEJ. Targeting the affective brain-a randomized controlled trial of real-time fMRI neurofeedback in patients with depression. Neuropsychopharmacology. 2018 Dec;43(13):2578-2585. doi: 10.1038/s41386-018-0126-5. Epub 2018 Jun 23. PMID 29967368
- [Background] Mehler DMA, Williams AN, Krause F, Luhrs M, Wise RG, Turner DL, Linden DEJ, Whittaker JR. The BOLD response in primary motor cortex and supplementary motor area during kinesthetic motor imagery based graded fMRI neurofeedback. Neuroimage. 2019 Jan 1;184:36-44. doi: 10.1016/j.neuroimage.2018.09.007. Epub 2018 Sep 8. PMID 30205210
- [Background] Paret C, Zaehringer J, Ruf M, Ende G, Schmahl C. The orbitofrontal cortex processes neurofeedback failure signals. Behav Brain Res. 2019 Sep 2;369:111938. doi: 10.1016/j.bbr.2019.111938. Epub 2019 May 6. PMID 31071348
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Sarasso E, Gardoni A, Zenere L, Canu E, Basaia S, Pelosin E, Volonte MA, Filippi M, Agosta F. Action observation and motor imagery improve motor imagery abilities in patients with Parkinson's disease - A functional MRI study. Parkinsonism Relat Disord. 2023 Nov;116:105858. doi: 10.1016/j.parkreldis.2023.105858. Epub 2023 Sep 22. PMID 37774517
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Skottnik L, Linden DEJ. Mental Imagery and Brain Regulation-New Links Between Psychotherapy and Neuroscience. Front Psychiatry. 2019 Oct 30;10:779. doi: 10.3389/fpsyt.2019.00779. eCollection 2019. PMID 31736799
- [Background] Skottnik L, Sorger B, Kamp T, Linden D, Goebel R. Success and failure of controlling the real-time functional magnetic resonance imaging neurofeedback signal are reflected in the striatum. Brain Behav. 2019 Mar;9(3):e01240. doi: 10.1002/brb3.1240. Epub 2019 Feb 20. PMID 30790474
- [Background] Subramanian L, Hindle JV, Johnston S, Roberts MV, Husain M, Goebel R, Linden D. Real-time functional magnetic resonance imaging neurofeedback for treatment of Parkinson's disease. J Neurosci. 2011 Nov 9;31(45):16309-17. doi: 10.1523/JNEUROSCI.3498-11.2011. PMID 22072682
- [Background] Subramanian L, Morris MB, Brosnan M, Turner DL, Morris HR, Linden DE. Functional Magnetic Resonance Imaging Neurofeedback-guided Motor Imagery Training and Motor Training for Parkinson's Disease: Randomized Trial. Front Behav Neurosci. 2016 Jun 8;10:111. doi: 10.3389/fnbeh.2016.00111. eCollection 2016. PMID 27375451
- [Background] Young KD, Siegle GJ, Zotev V, Phillips R, Misaki M, Yuan H, Drevets WC, Bodurka J. Randomized Clinical Trial of Real-Time fMRI Amygdala Neurofeedback for Major Depressive Disorder: Effects on Symptoms and Autobiographical Memory Recall. Am J Psychiatry. 2017 Aug 1;174(8):748-755. doi: 10.1176/appi.ajp.2017.16060637. Epub 2017 Apr 14. PMID 28407727
- [Background] Zahn R, Weingartner JH, Basilio R, Bado P, Mattos P, Sato JR, de Oliveira-Souza R, Fontenelle LF, Young AH, Moll J. Blame-rebalance fMRI neurofeedback in major depressive disorder: A randomised proof-of-concept trial. Neuroimage Clin. 2019;24:101992. doi: 10.1016/j.nicl.2019.101992. Epub 2019 Aug 25. PMID 31505367